CLINICAL TRIAL: NCT04936126
Title: Comparative Efficacy of Antidepressant Augmentation With Amantadine vs Pramipexole vs Quetiapine in Treatment-resistant Unipolar Depression: A Randomized Controlled Trial.
Brief Title: Comparison of Antidepressant Augmentation With Amantadine vs Pramipexole vs Quetiapine in Treatment Resistant Depression
Acronym: APQ-TRD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, BISWA RANJAN MISHRA, Additional Professor, Department of Psychiatry, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: T/EMF/Psych/19/49
Record Dates: First submitted 2021-06-14; First posted 2021-06-23 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Treatment Resistant Depression
Keywords: Treatment Resistant Depression; Augmentation; Amantadine; Pramipexole; BDNF; NGF
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Quetiapine Fumarate; Amantadine; Pramipexole

STUDY DESIGN:
Intervention Model Description: Prospective, parallel-arm, randomized, single-blind, controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will remain blind to the treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Quetiapine group (Active Comparator): Quetiapine XR 100 mg/day augmentation to the ongoing Sertraline treatment.
  Interventions: Drug: Quetiapine
- Amantadine group (Experimental): Amantadine 200 mg/day (in two divided doses) augmentation to the ongoing Sertraline treatment
  Interventions: Drug: Amantadine
- Pramipexole group (Experimental): Pramipexole 0.375 mg/day (in three divided doses) augmentation to the ongoing Sertraline treatment
  Interventions: Drug: Pramipexole

INTERVENTIONS:
Drug: Quetiapine — Quetiapine XR 100 mg/day augmentation to the ongoing Sertraline treatment for the study period
  Arms: Quetiapine group
Drug: Amantadine — Amantadine 200 mg/day (in two divided doses) augmentation to the ongoing Sertraline treatment for the study period
  Arms: Amantadine group
Drug: Pramipexole — Pramipexole 0.375 mg/day (in three divided doses) augmentation to the ongoing Sertraline treatment for the study period
  Arms: Pramipexole group

SUMMARY:
The present study has been designed to compare the efficacy and safety of augmentation of SSRIs with Amantadine vs Pramipexole vs the recommended Quetiapine augmentation in Treatment-Resistant Depression (TRD) and correlate the changes in depression scores with changes in the serum levels of Brain-derived neurotrophic factor (BDNF) and Nerve growth factor (NGF).

The proposed study will be a prospective, randomized, single-blind, controlled clinical trial in patients with TRD and will be conducted over a period of 2 years. The study cohort will comprise 150 patients with unipolar depression clinically diagnosed as TRD, who are currently on Sertraline treatment (dose range = 100-200 mg/day). At baseline, Hamilton Depression Scale (HAM-D 21 item) will be administered to determine the severity of depressive symptoms, Clinical Global Inventory (CGI) will be administered to determine the baseline severity of the illness. Serum BDNF, and NGF will be estimated by ELISA using commercially available Human ELISA kit. The sample will be divided into 3 equal treatment groups by block randomization technique, each group comprising of 50 patients.

Group 1 will receive Amantadine 200 mg/day (in two divided doses) augmentation to the ongoing Sertraline treatment. Group 2 will receive Pramipexole 0.375 mg/day (in three divided doses) augmentation to the ongoing Sertraline treatment. Group 3 will serve as the control arm and receive the recommended Quetiapine XR 100 mg/day augmentation to the ongoing Sertraline treatment.

The study cohort will be reassessed for the changes in HAM-D scores, CGI severity scores, Improvement score and Efficacy index, at 4 and 8 weeks follow up. The changes in Serum BDNF, and NGF will be estimated at the end of 8 weeks, to correlate with the change in severity of depressive symptoms. All the participants will be evaluated for any untoward side effects in a prescribed format for the Pharmacovigilance program of India (PVPI). The patient in either of the treatment arms, who are not responding to treatment or relapsing with aggravation of depressive symptoms will be switched on to Venlafaxine treatment or Electro-convulsive therapy (ECT) as decided by the treating team.

DETAILED DESCRIPTION:
STUDY OBJECTIVES:

Primary Objective

• To compare the change in the severity of symptoms of depression in terms of change in HAM-D scores between the treatment groups over 8 weeks.

Secondary Objective

* To compare the change in CGI scores between the treatment groups over 8 weeks.
* To evaluate the change in serum BDNF, serum NGF levels between the treatment groups over 8 weeks.
* To detect adverse drug reactions (if any) (prescribed format for Pharmacovigilance program of India PVPI)

Study design:

This study will be a hospital-based, prospective, randomized, single-blind, controlled clinical trial in patients with unipolar depression clinically diagnosed as TRD, which will be conducted over a period of 3 years.

Study population and eligibility:

The study cohort will comprise of 150 patients with the diagnosis of unipolar treatment-resistant depression (TRD), attending the in-patient or out-patient department of Psychiatry, All India Institute of Medical Sciences, Bhubaneswar. The patient should have received adequate trials of at least two antidepressants (one of which preferably should be an SSRI) at adequate dose and duration (> 6 weeks), with poor clinical response while on regular compliance. The patients fulfilling the criteria who are currently on Sertraline treatment (dose range = 100-200 mg/day), giving written informed consent will be recruited for the present study. The detailed history, relevant socio-demographic, and clinical data will be collected in a structured case record form (CRF).

Study Procedure and Data collection:

Baseline assessment:

At baseline, Hamilton Depression Scale (HAM-D 21 item) will be administered to determine the severity of depressive symptoms, Clinical Global Inventory (CGI) will be administered to determine the baseline severity of the illness. Serum BDNF, and NGF will be estimated by ELISA using commercially available Human ELISA kit.

Randomization:

The study cohort of 150 participants will be randomized into three treatment groups by block randomization technique (computer-generated) with 25 blocks, each block with 6 participants. The sample will be divided into 3 equal treatment groups, each group comprising of 50 patients.

Treatment Allocation:

Group 1 will receive Amantadine 200 mg/day (in two divided doses) augmentation to the ongoing Sertraline treatment. Group 2 will receive Pramipexole 0.375 mg/day (in three divided doses) augmentation to the ongoing Sertraline treatment. Group 3 will serve as the control arm and receive the recommended Quetiapine XR 100 mg/day augmentation to the ongoing Sertraline treatment.

Follow up assessment:

The study cohort will be reassessed for the changes in HAM-D scores, CGI severity scores, Improvement score, and Efficacy index, at 4 and 8 weeks follow up. The changes in Serum BDNF and NGF will be estimated at the end of 8 weeks, to correlate with the change in the severity of depressive symptoms.

Rescue Medication:

The patient in either of the treatment arms, who are not responding to treatment or relapsing with aggravation of depressive symptoms will be switched on to Venlafaxine treatment or ECT as decided by the treating team.

Safety evaluation:

All the participants will be evaluated for any untoward side effects like insomnia, restlessness, and agitation, etc. which will be documented and informed to the institutional ethics committee.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unipolar depression clinically diagnosed as TRD, who are currently on Sertraline treatment (dose range = 100-200 mg/day)
2. Patients aged 18-60 years of either sex

Exclusion Criteria:

1. Patients with Bipolar affective disorder
2. Patient with TRD on antidepressants other than Sertraline
3. History of psychoactive substance abuse or dependence
4. Co-morbid psychiatric, major medical, or neurological disorders
5. History of organicity or significant head injury
6. Pregnant and lactating women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-08-07 (Actual); Primary Completion 2024-07-07 (Estimated); Study Completion 2024-09-07 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Scale scores | 8 weeks
  Change in Hamilton Depression Scale scores 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression Higher scores indicating higher severity of depression

SECONDARY OUTCOMES:
Clinical Global Impression scores | 8 weeks
  Change in Clinical Global Impression scores CGI-S severity scores range from 1-7, with higher scores indicating greater severity of illness CGI-I Improvement score range from 1-7, with lower scores indicating improvement and higher scores indicating worsening
Serum Brain Derived Neurotrophic Factor | 8 weeks
  Change in Serum Brain Derived Neurotrophic Factor levels
Serum Nerve Growth Factor | 8 week
  Change in Serum Nerve Growth Factor
Rescue Medications | 8 weeks
  Number of patients in the Rescue medication group

CONTACTS AND LOCATIONS:
Overall Officials: Debadatta Mohapatra, MD, Study Chair — All India Institute of Medical Sciences, Bhubaneswar
Locations (1):
- All India Institute of Medical Sciences, Bhubaneswar, Odisha, India

REFERENCES:
- [Result] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Result] Kennedy SH, Giacobbe P. Treatment resistant depression--advances in somatic therapies. Ann Clin Psychiatry. 2007 Oct-Dec;19(4):279-87. doi: 10.1080/10401230701675222. PMID 18058285
- [Result] Fava M, Davidson KG. Definition and epidemiology of treatment-resistant depression. Psychiatr Clin North Am. 1996 Jun;19(2):179-200. doi: 10.1016/s0193-953x(05)70283-5. PMID 8827185
- [Result] Souery D, Amsterdam J, de Montigny C, Lecrubier Y, Montgomery S, Lipp O, Racagni G, Zohar J, Mendlewicz J. Treatment resistant depression: methodological overview and operational criteria. Eur Neuropsychopharmacol. 1999 Jan;9(1-2):83-91. doi: 10.1016/s0924-977x(98)00004-2. PMID 10082232
- [Result] Dold M, Kasper S. Evidence-based pharmacotherapy of treatment-resistant unipolar depression. Int J Psychiatry Clin Pract. 2017 Mar;21(1):13-23. doi: 10.1080/13651501.2016.1248852. Epub 2016 Nov 16. PMID 27848269
- [Result] Fleurence R, Williamson R, Jing Y, Kim E, Tran QV, Pikalov AS, Thase ME. A systematic review of augmentation strategies for patients with major depressive disorder. Psychopharmacol Bull. 2009;42(3):57-90. PMID 19752841
- [Derived] Mishra BR, Mohapatra D, Biswas T, Mishra A, Panigrahi S, Maiti R. Comparative efficacy of antidepressant augmentation with amantadine vs pramipexole in treatment-resistant unipolar depression: A randomised controlled trial. J Affect Disord. 2025 Dec 1;390:119891. doi: 10.1016/j.jad.2025.119891. Epub 2025 Jul 13. PMID 40659070